CLINICAL TRIAL: NCT00136812
Title: Treating Tobacco Dependence in Inpatient Psychiatry
Brief Title: Treating Tobacco Dependence in Inpatient Psychiatry - 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Judith Prochaska, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-18691-1; 5K23DA018691-05 (NIH)
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Results first posted 2016-03-23 (Estimated); Last update posted 2024-04-11 (Actual); Status verified 2024-03

CONDITIONS: Tobacco Use Cessation; Tobacco Use Disorder
Keywords: tobacco
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- enhanced usual care control (No Intervention): NRT during hospitalization with brief advice to stay quit once discharged
- stage-tailored intervention (Experimental): NRT during hospitalization with brief advice to stay quit once discharged plus a computer-delivered stage-tailored smoking cessation intervention with manual and counseling plus 10-weeks of nicotine patch available post-hospitalization
  Interventions: Behavioral: stage-tailored intervention

INTERVENTIONS:
Behavioral: stage-tailored intervention — This intervention consists of nicotine patch therapy during hospitalization; a stage-based self-help manual; an individualized, expert-system, feedback report at intake, 3 months and 6 months post-hospitalization with carbon copies sent to participants' outpatient clinicians; and an individual 30-min smoking cessation counseling sessions during hospitalization. Additionally, up to 10 weeks of nicotine patch is provided to intervention participants intending to stay quit following hospital discharge.
  Arms: stage-tailored intervention

SUMMARY:
The purpose of this study is to test in a randomized clinical trial a series of hypotheses concerning the efficacy of an extended expert-system intervention plus nicotine replacement therapy (NRT) for treating tobacco dependence among patients hospitalized on a smoke-free psychiatric unit.

DETAILED DESCRIPTION:
It is hypothesized that the intervention will be more effective than the enhanced standard care control condition (on-unit NRT with self-help brochure) in producing biochemically verified abstinence from cigarettes at 3-, 6-, 12-, and 18-months follow up. Additionally, intervention participants will exhibit greater stage progression, commitment to abstinence, and delay in relapse to smoking following hospital discharge, factors predictive of future success with quitting smoking. Smoking cessation treatments have been shown to be highly cost-effective with the general population of smokers, and cost is likely to be a consideration in efforts to incorporate additional services into an inpatient psychiatric setting. Therefore, a secondary specific aim is to model the cost-effectiveness of the smoking cessation intervention. Intervention efficacy will be examined in a university-based psychiatric inpatient unit. A smaller pilot study will examine translation of the intervention to a county hospital serving a more diversified patient population.

ELIGIBILITY:
Inclusion Criteria: Men and women over 18 years of age hospitalized on an inpatient psychiatric unit who report smoking at least 5 cigarettes per day; smoking at least 100 cigarettes in one's lifetime, residing in the San Francisco Bay Area with no plan to relocate outside of the area in the next 18 months, and access to a telephone for scheduling follow up assessments.

Exclusion Criteria: Dementia or other brain injury precluding ability to participate; non-English speaking; severe agitation, psychosis, or hostility; and medical contraindications to nicotine replacement therapy (NRT). Recruitment of acutely psychotic, manic, or hostile patients will be delayed until there is significant reduction of these symptoms. Medical contraindications are: myocardial infarction in the preceding 3 months, unstable angina pectoris, liver or kidney disease, current pregnancy or breast feeding, allergies to adhesives, or other medical conditions that the medical team deems incompatible with NRT use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2006-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Prochaska, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - San Francisco General Hospital, San Francisco, California
  - Langley Porter Psychiatric Institute, San Francisco, California

IPD SHARING:
Plan to Share IPD: No
no plan to make individual participant data available

REFERENCES:
- [Result] Barnett PG, Wong W, Jeffers A, Hall SM, Prochaska JJ. Cost-effectiveness of smoking cessation treatment initiated during psychiatric hospitalization: analysis from a randomized, controlled trial. J Clin Psychiatry. 2015 Oct;76(10):e1285-91. doi: 10.4088/JCP.14m09016. PMID 26528651

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult smokers (N=224) were recruited between July 2006 and December 2008 from the adult inpatient psychiatry unit at the Langley Porter Psychiatric Institute (LPPI) located on the University of California, San Francisco (UCSF) medical school campus.
Groups:
- Control: Usual care provided NRT during hospitalization with brief cessation advice.
- Brief Treatment: The intervention included a Transtheoretical Model-tailored computerized program and print workbook; brief on-unit counseling session; and nicotine replacement therapy (NRT) during hospitalization with access to 10 weeks of NRT post-hospitalization.
Period: Overall Study
Arm/Group | Control | Brief Treatment
Started | 111 | 113
Completed | 111 | 113
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Brief Treatment | Total
Number analyzed (Participants) | 111 | 113 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (14.1) | 39.9 (13.5) | 39.9 (14)
Sex/Gender, Customized [Number; unit: participants]
  Female | 71 | 63 | 134
  Male | 36 | 48 | 84
  Other | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: 7 Day Point Prevalence of Cigarette Abstinence
Time Frame: 3 mo, 6 mo, 12 mo, and 18 mo post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Brief Treatment
Number analyzed (Participants) | 111 | 113
Participants
  3 month | 3 | 14
  6 month | 6 | 14
  12 month | 10 | 18
  18 month | 7 | 18
Statistical Analysis 1: Comparison: Control vs Brief Treatment; To test the primary hypothesis, we ran a generalized estimating equation model with logit link function (PROC GENMOD in SAS version 9.2), to examine abstinence versus smoking status at the 3- through 18-month follow-ups by condition; Test type: Other — We used all available observations in a GEE analysis and did not impute missing data or drop observations; p = 0.018, generalized estimating equation model — P-value of <0.05 is considered statistically significant; Odds Ratio (OR) = 3.15, 95% CI 2-sided [1.22 to 8.14]

ADVERSE EVENTS:
Groups:
- 1: Enhanced Standard Care Control: enhanced standard care control
- 2: Intervention: intervention
  Tobacco Use Cessation: This intervention consists of nicotine patch therapy during hospitalization; a stage-based self-help manual; an individualized, expert-system, feedback report at intake, 3 months and 6 months post-hospitalization with carbon copies sent to participants' outpatient clinicians; and an individual 30-min smoking cessation counseling sessions during hospitalization. Additionally, up to 10 weeks of nicotine patch is provided to intervention participants intending to stay quit following hospital discharge.
Arm/Group | 1: Enhanced Standard Care Control | 2: Intervention
All-Cause Mortality (participants affected / at risk) | 2/111 | 2/113
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/113
Other Adverse Events (participants affected / at risk) | 0/111 | 0/113

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No